CLINICAL TRIAL: NCT04191278
Title: Mobile Health Interventions for Varenicline Adherence Among HIV-positive Smokers
Brief Title: Mobile Health Interventions for Medication Adherence Among PLWH
Acronym: HIVSMART
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID prevented study initiation
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100107; K01DA043413 (NIH)
Record Dates: First submitted 2019-11-27; First posted 2019-12-09 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-09

CONDITIONS: HIV/AIDS; Smoking; Smoking Cessation; HIV
Keywords: Smoking; mHealth; Chantix; Varenicline; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three study conditions: 1) varenicline alone; 2) varenicline + mobile health app; 3) varenicline + mobile health app + contingency management
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Varenicline (Active Comparator): An α4β2 nicotinic acetylcholine receptor partial agonist
  Interventions: Drug: Varenicline
- Varenicline + mobile app (Experimental): An α4β2 nicotinic acetylcholine receptor partial agonist + a mobile phone application designed to improve adherence to medications
  Interventions: Drug: Varenicline; Device: Mobile phone application
- Varenicline + mobile app + contingency management (Experimental): An α4β2 nicotinic acetylcholine receptor partial agonist + a mobile phone application designed to improve adherence to medications + monetary reinforcers for being adherent to medication
  Interventions: Drug: Varenicline; Device: Mobile phone application; Behavioral: Contingency management

INTERVENTIONS:
Drug: Varenicline — All participants will receive a standard 12-week course of varenicline tartrate. Participants will receive 0.5 mg tablets per oral (PO) once daily for days 1-3, 0.5 mg tablets PO twice daily for days 4-7, and 1 mg tablets PO twice daily for days 8-84
  Other Names: Chantix
Device: Mobile phone application — Participants randomized to 2 of the 3 study groups will receive a mobile phone application designed to improve adherence to medication. The app has a number of functions, including: a) reminders to take medication; b) information about coping strategies for dealing with side effects and withdrawal symptoms; c) provision of a personalized graphical display of treatment progress (e.g., adherence, side effects); d) camera-based verification of having taken medication.
  Arms: Varenicline + mobile app; Varenicline + mobile app + contingency management
Behavioral: Contingency management — Participants randomized to 1 of the 3 study groups will receive monetary reinforcement contingent upon verified medication adherence behaviors. Participants in the other 2 groups will be yoked to a participant in the CM group so that they also have a chance of earning monetary reinforcers, though not contingent upon their own behaviors.
  Arms: Varenicline + mobile app + contingency management

SUMMARY:
Cigarette smoking remains highly prevalent among persons living with HIV (PLWH). Quitting smoking can have important health benefits for this population. However, PLWH have historically had a difficult time quitting smoking. This is likely due, at least in part, to poor medication adherence.

Poor adherence to medication is a well-documented issue among PLWH. Research shows that not taking smoking cessation medications as prescribed can limit their treatment effectiveness. Improving adherence to smoking cessation medications will likely increase smoking cessation attempt success.

Mobile phone applications and behavioral interventions show promise for improving adherence to smoking cessation medications and cessation outcomes among PLWH. Therefore, this trial will assess 1) whether a mobile phone application is a feasible and acceptable intervention for improving medication adherence; 2) whether use of the mobile phone app improves adherence to varenicline; and 3) smoking cessation outcomes.

DETAILED DESCRIPTION:
Cigarette smoking is a significant public health problem among persons living with HIV (PLWH). The prevalence of smoking among PLWH is 40-75%, compared to approximately 15% in the general population. In PLWH, smoking confers increased risk of cardiovascular disease, respiratory conditions, lung cancer, poor adherence to antiretroviral (ARV) therapy, poor HIV treatment outcomes, and all-cause mortality. Approximately 24% of deaths among PWLH on ARV are attributable to tobacco use. Moreover, smokers with HIV lose more life years to smoking than to HIV itself (13 versus 5 years).

Smoking cessation is a challenge for smokers with HIV. Smokers with HIV are interested in quitting, yet most quit attempts end in relapse. Poor cessation outcomes are likely attributable, in part, to poor adherence to smoking cessation medications. Not taking varenicline as prescribed significantly limits treatment effectiveness. Adherence to varenicline in smokers with HIV is poor, with only 56-62% of individuals in clinical trials taking the medication as prescribed. Putatively, real world adherence is expected to be lower. Medication adherence is a well-documented issue in HIV: only 62% achieve optimal adherence to ARV. Interventions are needed to improve smoking cessation medication adherence among smokers with HIV. Such interventions will improve cessation and reduce the burden of smoking in this population.

Mobile phone-delivered interventions show promise for improving cessation outcomes in smokers living with HIV. However, an intervention that provided text message medication reminders and motivational cessation messages with or without phone-delivered counseling, as compared to a control group, yielded no group differences for varenicline adherence. Thus, it is possible that more intensive, and multi-component, interventions are required to improve the effectiveness of mobile-phone-based interventions.

This trial will: 1) assess the feasibility and acceptability of a mobile phone app that aims to increase medication adherence; 2) whether use of the app and/or contingency management increases adherence to varenicline over varenicline treatment as usual; and 3) monitor smoking cessation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* HIV-positive
* Currently engaged with an HIV care provider
* Interested in quitting smoking within the next 30 days
* Has an Android (v5.x.x or Lollipop) or iOS (v6.0) smartphone (interested participants without a compatible smartphone will be provided one, with costs offset by the study team)
* English-speaking
* Capable of giving written informed consent

Exclusion Criteria:

* Inability to attend study sessions
* Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator, Study Physician, and/or participant's HIV care provider
* Current use of nicotine replacement therapy or other smoking cessation treatment (e.g., bupropion)
* Pregnant, planning to become pregnant, nursing, or becoming pregnant during the study
* BAL >0.000 at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The average number of times per day that participants initiate an interaction with mobile app | Daily throughout study duration (12 weeks)
  The average number of times per day that participants initiate an interaction with the app, as measured by background analytics
The average number of times per day participants respond to a prompt from mobile app | Daily throughout study duration (12 weeks)
  The average number of times per day that participants respond to prompts from the app, as measured by background analytics
Technical issues with using the mobile app | Weekly throughout study (once every week for 12 weeks)
  Average number of technical issues reported by participants throughout the course of the study
Perceived usefulness of mSMART app | Week 12
  Participants will be asked to respond to the following: "Overall, I find the mSMART app useful for remembering to take my varenicline." Response options include: Strongly disagree; Somewhat disagree; neither agree nor disagree; somewhat agree; strongly agree.
Perceived ease of use of mSMART app | Week 12
  Participants will be asked to respond to the following: "Overall, I find the mSMART app easy to use." Response options include: Strongly disagree; Somewhat disagree; neither agree nor disagree; somewhat agree; strongly agree.

SECONDARY OUTCOMES:
Adherence to varenicline | Weekly throughout study duration (once a week, over the course of 12 weeks)
  Percentage of varenicline pills taken as directed, as measured via pill counts
Concentration of expired breath carbon monoxide | Baseline and Weekly throughout study (once every week for 12 weeks)
  Participants will provide an expired breath carbon monoxide sample at each study visit, measured in parts per million. Smoking cessation will be defined as a measured carbon monoxide sample that is ≤50% lower than their expired breath carbon monoxide that was measured at baseline
Concentration of cotinine in urine sample | Weekly throughout study (once every week for 12 weeks)
  Participants will provide a urine sample at each study visit. These samples will be tested with a rapid urinary cotinine strip that indicates whether or not the participant has been abstinent from smoking (measured in ng of cotinine per mL of urine).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren R Pacek, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No